CLINICAL TRIAL: NCT00984685
Title: "Assessment of Risk Factors for Depression Treatment at a Safety Net Clinic"
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Scranton-Temple Residency Program (Other)
Responsible Party: Dr. John R Guzek MD, Scranton-Temple Residency Program
Other Study IDs: STRP0002
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- depression: Patients diagnosed with depression before April 15, 2009

SUMMARY:
The purpose of the study is to identify the barriers for effective treatment of depression, specifically whether modified CHIS Scale is a valid tool for identifying the high risk patients for depression.

DETAILED DESCRIPTION:
Depression is a major illness that affects 10% of the population in a medical setting. It is often under diagnosed and under treated. It is an illness that can challenge a persons ability to perform even routine daily activities. Review of the charts of patients diagnosed with depression showed 80% of the patients do not have follow up appointments. We wondered if modified CHIS scale could identify the risk factors for medication non-adherence.

We hypothesised that modified CHIS Scale an effective tool ,for identifying the compliance of patients with the antidepressant medication.

We are conducting a retrospective cohort study at two of our residency based clinics by interviewing approximately 100 patients with CHIS Scale and PHQ9 Questionnaire on their office visits

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of depression before April 15, 2009
* At least one visit since April 15, 2008
* Age 18+

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with the diagnosis of depression in theprimary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-08; Primary Completion 2009-09 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
proportion of anti-depressant prescriptions filled | August 1, 2008 through July 31, 2009

CONTACTS AND LOCATIONS:
Overall Officials: John R Guzek, MD, Principal Investigator — Scranton-Temple Residency Program
Locations (1):
- Scranton Temple Residency Program, Scranton, Pennsylvania, United States